CLINICAL TRIAL: NCT01738828
Title: Genetic Loci and the Burden of Atherosclerotic Lesions
Brief Title: GLOBAL Clinical Study
Acronym: GLOBAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Global Genomics Group, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR0001
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, buffy coat and RNA PAXgene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with CAD
- Subjects without CAD

SUMMARY:
The GLOBAL study is an international multi-center, prospective study designed to enroll up to 10,000 consecutive eligible subjects who are clinically referred for coronary CT angiography for assessment of suspected coronary artery disease (CAD).

The purpose of the study is to perform extensive biomarker analysis of atherosclerosis in patients phenotyped using advanced imaging modalities of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-90
2. Caucasian and of Non-Hispanic or Non-Latino origin
3. Referral for coronary CT angiography to evaluate for presence of CAD
4. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form

Exclusion Criteria:

1. Immunosuppressive or immunomodulatory therapy including any dose of systemic corticosteroids in the preceding 30 days (except if steroids are administered as pre-medication prior to contrast administration for CT scan within 24 hours).
2. Chemotherapy in the preceding year
3. Major surgery in the preceding 2 months
4. Blood or blood product transfusion in the preceding 2 months
5. Subjects for whom coronary CT angiography is contraindicated per institutional standard of care
6. Subjects with previous coronary arterial revascularization (PCI or CABG)
7. Subjects with atrial fibrillation/flutter or frequent irregular or rapid heart rhythms, which occurred within the past 3 months
8. Subjects with a pacemaker or implantable cardioverter-defibrillator implant
9. Active congestive heart failure or the presence of known non-ischemic cardiomyopathy
10. Known genetic disorders of atherosclerosis, lipid or lipoprotein metabolism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for clinically indicated coronary CT angiography for an assessment of possible CAD are potential study candidates.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Genome-Wide Association | Baseline
  The primary analysis will be a genome-wide association analysis, to determine candidate genes and markers underlying coronary artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Szilard Voros, MD, Study Director — Global Genomics Group, LLC
Locations (48):
- United States (29):
  - Heart Center Research, Huntsville, Alabama
  - The University of Arizona, Tucson, Arizona
  - Sutter Roseville Medical Center, Roseville, California
  - Colorado Health Medical Group, Colorado Springs, Colorado
  - The MedStar Heart Research Institute, Washington D.C., District of Columbia
  - Elite Research and Clinical Trials, Miami Beach, Florida
  - Georgia Regents University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - United Heart and Vascular Center, Saint Paul, Minnesota
  - Midwest Heart and Vascular Specialists, Kansas City, Missouri
  - Saint Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Long Island Heart Associates, Mineloa, New York
  - St. Francis Hospital, Roslyn, New York
  - Zwanger Pesiri Radiology, Stony Brook, New York
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - The Linder Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Berks Cardiologists, Wyomissing, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Cardiac Study Center, Puyallup, Washington
- Australia (6):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Monash Heart, Clayton, Victoria
  - Alfred Hospital, Melbourne, Victoria
- The University of British Columbia, Vancouver, British Columbia, Canada
- Poliklinika Sunce, Zagreb, Croatia
- Germany (2):
  - University of Erlangen, Erlangen
  - Isar Heart Center, Munich
- Hungary (2):
  - Semmelweis University, Budapest
  - University of Kaposvar, Kaposvár
- Netherlands (2):
  - Meander Medical Center, Amersfoot
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
- Institute of Cardiology, Warsaw, Poland
- United Kingdom (4):
  - Ulster Hospital, Belfast
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - Plymouth Hospitals NHS Trust of Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Drobni ZD, Kolossvary M, Karady J, Jermendy AL, Tarnoki AD, Tarnoki DL, Simon J, Szilveszter B, Littvay L, Voros S, Jermendy G, Merkely B, Maurovich-Horvat P. Heritability of Coronary Artery Disease: Insights From a Classical Twin Study. Circ Cardiovasc Imaging. 2022 Mar;15(3):e013348. doi: 10.1161/CIRCIMAGING.121.013348. Epub 2022 Mar 15. PMID 35290075
- [Derived] Whitaker J, Karady J, Karim R, Tobon-Gomez C, Fastl T, Razeghi O, O'Neill L, Decroocq M, Williams S, Corrado C, Mukherjee RK, Sim I, O'Hare D, Kotadia I, Kolossvary M, Merkely B, Littvay L, Tarnoki AD, Tarnoki DL, Voros S, Razavi R, O'Neill M, Rajani R, Maurovich Horvat P, Niederer S. Standardised computed tomographic assessment of left atrial morphology and tissue thickness in humans. Int J Cardiol Heart Vasc. 2020 Dec 24;32:100694. doi: 10.1016/j.ijcha.2020.100694. eCollection 2021 Feb. PMID 33392384
- [Derived] Voros S, Maurovich-Horvat P, Marvasty IB, Bansal AT, Barnes MR, Vazquez G, Murray SS, Voros V, Merkely B, Brown BO, Warnick GR. Precision phenotyping, panomics, and system-level bioinformatics to delineate complex biologies of atherosclerosis: rationale and design of the "Genetic Loci and the Burden of Atherosclerotic Lesions" study. J Cardiovasc Comput Tomogr. 2014 Nov-Dec;8(6):442-51. doi: 10.1016/j.jcct.2014.08.006. Epub 2014 Sep 6. PMID 25439791